CLINICAL TRIAL: NCT07285668
Title: Phase I Study of Prophylactic TCRαβ+ and CD19+ Depleted Donor Lymphocyte Infusion After Allogeneic Stem Cell Transplant in High-Risk Patients With Hematologic Malignancies
Brief Title: Prophylactic TCRaB+ and CD19+ Depleted Donor Lymphocyte Infusion After Allogeneic Stem Cell Transplant in High-Risk Patients With Hematologic Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1405; UW25034 (Other: OnCore ID); Protocol Version 8/8/25 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancies
Keywords: allogeneic donor; Lymphocyte Infusion
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-center, phase I 3x3 dose-escalation study with expansion cohort, open label, non-randomized, non-placebo controlled, single-group assignment study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Dose Escalation Cohort Level 1 (Experimental): 1 x 10^6 CD3-CD56+/kg
  Interventions: Device: Allogeneic donor TCRαβ+/CD19+ cell-depleted peripheral blood mononuclear cells
- Dose Escalation Cohort Level 2 (Experimental): 2 X 10^6 CD3-CD56+/kg
  Interventions: Device: Allogeneic donor TCRαβ+/CD19+ cell-depleted peripheral blood mononuclear cells
- Dose Escalation Cohort Level 3 (Experimental): 5 X 10^6 CD3-CD56+/kg
  Interventions: Device: Allogeneic donor TCRαβ+/CD19+ cell-depleted peripheral blood mononuclear cells
- Dose Escalation Cohort Level -1 (Experimental): 0.5 x 10^6 CD3-CD56+/kg
  Dose to be used only if Dose Level 1 is not tolerated.
  Interventions: Device: Allogeneic donor TCRαβ+/CD19+ cell-depleted peripheral blood mononuclear cells

INTERVENTIONS:
Device: Allogeneic donor TCRαβ+/CD19+ cell-depleted peripheral blood mononuclear cells — Single intravenous dose of allogeneic donor TCRαβ+/CD19+ cell-depleted peripheral blood mononuclear cells (i.e., αβT/B dep-DLI), where the dose is based on the natural killer (NK) cell (CD3-CD56+) content in the DLI product. Each participant will receive one of four DLI doses depending upon cohort to which the participant is enrolled.

SUMMARY:
This study is being done to assess the safety and determine the maximum tolerable dose (MTD) of TCRαβ+/CD19+-depleted Donor Lymphocyte Infusion (αβT/B dep-DLI) after allogeneic stem cell transplant (allo-SCT) in highrisk patients with hematologic malignancies.

DETAILED DESCRIPTION:
Primary Objectives

* To assess safety of prophylactic TCRαβ+/CD19+ depleted donor lymphocyte infusion (αβT/B dep-DLI) after allogeneic stem cell transplant (allo-SCT) in high-risk patients with hematologic malignancies
* To determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) of αβT/B dep-DLI

Secondary Objectives

* To assess the feasibility of αβT/B dep-DLI
* To assess additional safety parameters after αβT/B dep-DLI
* To assess the efficacy of αβT/B dep-DLI

For the dose escalation phase: Maximum Tolerated Dose (MTD) and Maximum Administered Dose (MAD) is defined as the highest dose level where less than 2 of 6 participants experience a dose limiting toxicity (DLT).

Each dose level will be followed for DLTs until day 28 post donor lymphocyte infusion (DLI). Starting at dose level 1:

* If 0 of 3 participants experiences DLT, increase to next dose level for next 3 participants.
* If 1 of 3 participants experience DLT, enroll 3 participants at same dose level.

  * If no additional DLTs (1 of 6), move on to next dose level.
  * If 2 of 6 participants experience DLT, enroll 3 participants into lower dose level.
* If 0 or 1 participants experience DLT at lower level, this will be the MTD.

Once the MTD or MAD is determined, an expansion cohort will be enrolled into that dose level.

All participants will be followed for 2 years after DLI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-risk myeloid or lymphoid malignancies determined to be eligible to undergo a related, allo-SCT using Disease Risk Index (DRI), including the conditions listed below. These criteria apply BEFORE cyto-reductive therapy given within 28 days of planned conditioning:

  * Refractory acute myelogenous or lymphoid leukemia
  * Relapsed acute myelogenous or lymphoid leukemia
  * Myelodysplastic syndromes with 5 percent or more blasts
  * Chronic myelogenous leukemia in chronic phase 3 or more, blast phase presently, or second accelerated phase
  * Recurrent or refractory malignant lymphoma or Hodgkin's disease with less than a partial response at transplant
  * High risk chronic lymphocytic leukemia defined as no response or stable disease to the most recent treatment regimen
  * Other high risk hematologic malignancies for which allo-SCT is deemed clinically necessary per PI and based on institutional standards
* The donor for the allo-SCT will have been identified prior to participant recruitment and must be:

  * Related AND
  * Matched OR mismatched OR haploidentical at Human Leukocyte Antigen (HLA) HLA-A, -B, -C, and -DRB1 by molecular methods
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
* Ability to understand and willingness to sign written informed consent document
* Willing to comply with all study procedures and be available for the duration of the study
* Individuals in sexual relationships that could result in pregnancy or impregnation of their partner must use an acceptable method of contraception§ from enrollment until 4 weeks after completing study treatment.

Exclusion Criteria:

* Poor organ function as follows (According to the pre-transplant workups results):

  * Creatinine greater than or equal to 2.0 mg/dL
  * Serum Glutamic Oxaloacetic Transaminase (SGOT) and Serum Glutamic Pyruvic Transaminase (SGPT) greater than or equal to 5 x Upper Limit of Normal (ULN). Liver biopsy preferred for such patients.
  * Bilirubin greater than or equal to 3 x ULN (unless Gilbert's syndrome)
  * Diffusing capacity of the Lungs for Carbon Monoxide (DLCO) less than 50 percent corrected for hemoglobin
  * Left ventricular ejection fraction or shortening fraction less than 40 percent

NOTE: Exceptions to the above organ function exclusion criteria are allowable only with assent of the PI since the risks and benefits must be addressed for patients with potentially incurable hematologic malignancies. Such exceptions will be clearly documented in the subject's research record and will not be considered a deviation.

* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) from DLI to day 28 post-DLI | up to day 28 post-DLI (approximately day 63 on study)
  To assess safety of prophylactic TCRαβ+/CD19+ depleted donor lymphocyte infusion (αβT/B dep-DLI) after allogeneic stem cell transplant (allo-SCT) in high-risk patients with hematologic malignancies, incidence of AEs will be reported.
Maximum Tolerated Dose or Maximum Administered Dose | up to day 28 post-DLI (approximately day 63 on study)
  MTD/MAD defined as the highest dose level at which less than 2 of 6 participants experience a DLT.

SECONDARY OUTCOMES:
Incidence of grade II-IV acute Graft-versus-Host Disease (aGVHD) after αβT/B dep-DLI | up to day 28 post-DLI (approximately day 63 on study)
  To assess additional safety parameters after allo-SCT in high-risk patients with hematologic malignancies, Incidence of grade II-IV aGVHD after αβT/B dep-DLI will be reported.
Cumulative incidence of severe grade III-IV aGVHD after αβT/B dep-DLI | up to day 28 post-DLI (approximately day 63 on study)
  To assess additional safety parameters after allo-SCT in high-risk patients with hematologic malignancies, cumulative incidence of severe grade III-IV aGVHD after αβT/B dep-DLI will be reported.
Chronic Graft-versus-Host Disease (GVHD) incidence after αβT/B dep-DLI | up to day 28 post-DLI (approximately day 63 on study)
  To assess additional safety parameters after allo-SCT in high-risk patients with hematologic malignancies, chronic GVHD incidence after αβT/B dep-DLI will be reported.
Efficacy assessed by 1 year Progression Free Survival (PFS) | up to 1 year
  To assess the efficacy of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, 1 year PFS will be reported.
Efficacy Assessed by Non-Relapse Mortality | up to 2 years
  To assess the efficacy of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, non-relapse mortality will be reported.
Efficacy Assessed by Overall Survival | up to 2 years
  To assess the efficacy of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, overall survival will be reported.
Efficacy Assessed by Incidence of Cytomegalovirus (CMV) Reactivation | up to 2 years
  To assess the efficacy of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, incidence of CMV Reactivation will be reported.
Efficacy Assessed by Incidence of Fungal Infection | up to 2 years
  To assess the efficacy of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, incidence of fungal infections will be reported.
Efficacy Assessed by Incidence of Full Chimerism (CD3 compartment) | up to 2 years
  To assess the efficacy of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, incidence of full chimerism will be reported.
Efficacy Assessed by Immunoglobulin Levels | up to 2 years
  To assess the efficacy of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, quantitative immunoglobulin levels will be reported.
Efficacy Assessed by Lymphocyte Panel Analysis | up to 2 years
  To assess the efficacy of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, lymphocyte subset panel analysis will be conducted and reported.
Feasibility assessed by percentage of enrolled participants who are able to receive depleted DLI | up to approximately 35 days
  To assess the feasibility of prophylactic αβT/B dep-DLI after allo-SCT in high-risk patients with hematologic malignancies, the percentage of enrolled participants who are able to receive depleted DLI will be reported.

OTHER OUTCOMES:
Number of regulatory T cells | up to 2 years
  To assess the effect of regulatory T cells on safety and efficacy of prophylactic αβT/B dep-DLI following allo-SCT in high-risk patients with hematologic malignancies, enumeration of regulatory T cells by flow analysis of peripheral blood mononuclear cells (PBMC) using combinations of monoclonal antibodies specific for CD4, CD25, FoxP3 or CD127 will be completed and reported.
Measurable Residual Disease (MRD) | up to 2 years
  Flow cytometry will be used to assess the efficacy of αβT/B dep-DLI in eliminating MRD in patients with myeloid leukemia or Myelodysplastic Syndrome (MDS). Flow cytometry or ClonoSeq will be used for Acute Lymphoblastic Leukemia (ALL) or Chronic Lymphocytic Leukemia (CLL).

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Galipeau, MD, FRCP(C), Study Director — UW School of Medicine and Public Health; Hongtao Liu, MD, PhD, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The Principal Investigator, Sponsor and funding institutions (if applicable) will ensure that all mechanisms used to share data include proper plans and safeguards to protect the rights and privacy of participants who participate in this research. Data from this study may be requested from other researchers 5 years after the completion of the primary endpoint by contacting the Principal Investigator, Dr. Hongtao Liu.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 5 years after the completion of the primary endpoint

REFERENCES:
- See also: Stem Cell and Regenerative Medicine Center — https://stemcells.wisc.edu/staff/galipeau-jacques/